CLINICAL TRIAL: NCT05608954
Title: Effects of Physical Therapy on the Multisystems of Children With Cerebral Palsy: a Longitudinal Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Professor, Federal University of Health Science of Porto Alegre
Other Study IDs: Cerebral Palsy longitudinal
Record Dates: First submitted 2022-02-05; First posted 2022-11-08 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy; Physical Therapy Modalities
Keywords: Cerebral Palsy; Physical Therapy Modalities; Longitudinal Studies; Disabled Children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical Therapy Modalities: Children diagnosed with cerebral palsy will be followed longitudinally in their therapies within the physiotherapeutic treatment.
  Interventions: Other: Bobath Concept; Other: Pediasuit; Other: Locomotor training; Other: Stretching; Other: Psychomotricity; Other: Virtual reality

INTERVENTIONS:
Other: Bobath Concept — Handling of the Bobath Concept
Other: Pediasuit — Pediasuit
Other: Locomotor training — Locomotor training
Other: Stretching — Active, passive, active-assisted stretching
Other: Psychomotricity — Psychomotor skills
Other: Virtual reality — Virtual reality

SUMMARY:
Cerebral Palsy (CP) refers to childhood movement and posture disorders, whose severity, patterns of motor involvement and associated impairments are very varied. It is the most prevalent type of physical disability in children. Any non-progressive central nervous system (CNS) lesion that occurs in the prenatal, perinatal and postnatal period up to 2 years of life is considered CP. Thus, the present work aims to evaluate, monitor and verify the effects of physical therapy interventions on gross motor function, spasticity, balance, muscle activation, fatigue, respiratory system, functionality and social participation in children with cerebral palsy. This work will use some evaluation scales such as the Gross Motor Function Measure (GMFM-66), the Modified Ashworth Scale (MAS), the Early Clinical Assessment of Balance (ECAB), electromyography, the Fatigue Severity Scale and the Pediatric Functional Status. Scale. In addition to questionnaires, which will be applied directly to parents/caregivers, such as the Young Children's Participation and Environment Measure (YC-PEM), the PEDI (Pediatric Evaluation Disability Inventory) and the Goal Attainment Scaling (GAS).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Cerebral Palsy
* aged between 0-12 years
* classified in all the levels of the GMFCS
* those responsible agree to release the minor to participate in the study and sign the Free and Informed Consent Form (FICT)

Exclusion Criteria:

* have had botulinum toxin applied 6 months before the intervention
* recent surgery
* other physical abnormalities, genetic or severe syndromes.

Ages: 0 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 0 to 12 years old, diagnosed with cerebral palsy
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function | 1 year
  Measurement of Gross Motor Function
Gross Motor Function Classification System | Levels I - V. Higher scores mean a worse outcome
  Scale Gross Motor Function Classification System

SECONDARY OUTCOMES:
Electromyography | 1 year
  Muscle activation
Early Clinical Assessment of Balance - ECAB | 1 year
  Postural control and balance
Modified Ashworth Scale (MAS) | 1 year
  Muscle tone
Fatigue Severity Scale | 1 year
  Muscle fatigue
Pediatric Functional Status Scale | 1 year
  Functional status
YC-PEM - Young Children's Participation and Environment Measure | 1 year
  Level of participation and qualities of the environment in which these activities take place.
PEDI (Pediatric Evaluation Disability Inventory) | 1 year
  Detailed description of the child's functional performance, documenting its longitudinal changes in three functional areas: self-care, mobility and social function.
GAS (Goal Attainment Scaling) | 1 year
  Evaluation of results obtained in family therapy, or in an intervention program

CONTACTS AND LOCATIONS:
Overall Officials: Franciele Zardo, Msc, Principal Investigator — UFCSPA: Universidade Federal de Ciencias da Saude de Porto Alegre
Locations (1):
- Franciele Zardo, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No